CLINICAL TRIAL: NCT00920400
Title: Value of Fecal Calprotectin in Upper Gastrointestinal Disease
Brief Title: Diagnostic Value of Fecal Calprotectin in Disorders of the Upper Gastrointestinal Tract
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Professor Christoph Beglinger, Head of Gastroenterology & Hepatology, University Hospital Basel
Other Study IDs: CALPROTECT
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Peptic Esophagitis; Peptic Ulcer; Functional Dyspepsia; Irritable Bowel Syndrome; Inflammatory Bowel Diseases
MeSH Terms: conditions — Esophagitis, Peptic; Peptic Ulcer; Irritable Bowel Syndrome; Inflammatory Bowel Diseases

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy samples (stomach, duodenum) will be stored by the Department of Pathology at the University Hospital Basel
Oversight: Data Monitoring Committee: No

SUMMARY:
Fecal calprotectin is a very sensitive non-invasive inflammation marker in the detection of inflammatory bowel disease and, to a lesser degree, has also proven to be useful in adenomatous polyps, neoplasias, and infectious gastroenteritis. Elevated calprotectin levels can also be found in patients with lesion only in the upper gastrointestinal tract. However, the diagnostic value of calprotectin has never been tested in this setting. The aim of the study is therefore to determine the diagnostic value of fecal calprotectin in patients with diseases of the upper gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for upper gastrointestinal endoscopy for any reason
* Older than 18 years

Exclusion Criteria:

* Patients who are not able to provide informed consent
* Patients who are not able to provide a stool sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 consecutive patients undergoing upper endoscopy at the Department of Gastroenterology & Hepatology at the University Hospital Basel
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Department of Gastroenterology & Hepatology, Basel, Basel-Stand, Switzerland